CLINICAL TRIAL: NCT05075850
Title: PatiEnt Neuropsychological outcomeS After laseR Ablation
Acronym: PENSAR
Status: Completed | Type: Observational
Sponsor: Monteris Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: PENSAR LAANTERN Registry
Record Dates: First submitted 2021-09-15; First posted 2021-10-13 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Change
Keywords: Quality of Life; Neuropsychological Test Scores; Visual Field

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Neuroblate System — All subjects will undergo comprehensive neuropsychological assessment post-LITT per standard of care practice.
  Visual field testing will be conducted in a subset of enrolled patients.

SUMMARY:
PatiEnt Neuropsychological outcomeS After laseR ablation

DETAILED DESCRIPTION:
This is a multicenter sub-study that will include comprehensive neuropsychological assessment data collection done at baseline (within 1 year prior to the index LITT procedure) and at follow-up (at least 6 months from the index LITT procedure). Visual field testing will be conducted in a subset of enrolled patients. Up to 250 subjects may be enrolled at up to 15 study sites.

ELIGIBILITY:
Inclusion Criteria:

1. Patient or legally authorized representative provides written authorization and/or consent.
2. Patient is enrolled in the LAANTERN trial and had an epilepsy diagnosis without the presence of a malignant brain tumor.
3. Patient is 16 years of age or older.
4. Patient has completed a baseline comprehensive neuropsychological assessment with a neuropsychologist.

Exclusion Criteria:

1. Patient does not complete the index LITT procedure as specified in the LAANTERN registry.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study is being conducted as a sub-study within the LAANTERN registry; therefore, all enrolled patients in PENSAR must be consented to both protocols.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Landazuri, MD, Principal Investigator — University of Kansas
Locations (7):
- United States (7):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Advent Health Orlando, Orlando, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- PENSAR Subjects: All eligible study subjects who underwent LITT with the NeuroBlate System and completed study-related testing.
Period: Overall Study
Arm/Group | PENSAR Subjects
Started | 81
Completed | 47
Not Completed | 34
Not completed — Did not completed follow-up questionnaires | 34

BASELINE CHARACTERISTICS:
Population: 47 subjects completed baseline PENSAR study testing.
Arm/Group | PENSAR Subjects
Number analyzed (Participants) | 47
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 38.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 42
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Site-determined Cognitive Changes Per Domain
Description: Neuropsychological test data collected will describe cognitive domain specific changes as a cohort. Change will be assessed from raw test scores and demographically corrected standardized scores (where available). For this study, collected cognitive domains include Language (Boston Naming Test), Executive Function (Trails Making Test), Attention (Wechsler Adult Intelligence Scale 3 Digital Span Test), Verbal Memory (Logical Memory Test), Visual Memory (Brief Visiospacial Memory Test), Verbal Fluency (Animal Fluency Test), and Motor Function (Grooved Pegboard Test).
Time Frame: At least six months from baseline assessment. Subjects were analyzed even if they only had 1 test performed. The baseline test information can still be used even if they didn't have follow up testing done.
Population: Subjects who had LITT and completed baseline and follow-up testing.
Measure: Mean (Standard Deviation); unit: Score
Groups:
- PENSAR Subjects Baseline: All eligible study subjects who underwent LITT with the NeuroBlate System and completed Baseline study related testing
- PENSAR Subjects Follow-Up: All eligible study subjects who underwent LITT with the NeuroBlate System and completed Follow-Up study related testing
Arm/Group | PENSAR Subjects Baseline | PENSAR Subjects Follow-Up
Number analyzed (Participants) | 47 | 47
Score
  Boston Naming (range 13-60. Higher score is better): number analyzed (Participants) | 31 | 34
  Boston Naming (range 13-60. Higher score is better) | 49 (9.7) | 50.7 (6.6)
  Trails Making (range 16-291. Higher value is worse): number analyzed (Participants) | 36 | 40
  Trails Making (range 16-291. Higher value is worse) | 32.9 (15.4) | 35.3 (27.7)
  Wechsler Adult Intelligence Scale 3 Digital Span (range 2-58. Lower score is better): number analyzed (Participants) | 38 | 38
  Wechsler Adult Intelligence Scale 3 Digital Span (range 2-58. Lower score is better) | 13.1 (6.1) | 14.6 (9.8)
  Logical Memory (range 0-32. Higher score is better): number analyzed (Participants) | 19 | 32
  Logical Memory (range 0-32. Higher score is better) | 22.3 (6.0) | 18.9 (6.5)
  Brief Visuospacial Memory Test (range 0-33. Higher score is better): number analyzed (Participants) | 35 | 36
  Brief Visuospacial Memory Test (range 0-33. Higher score is better) | 20.1 (7.3) | 18.8 (8.3)
  Animal Fluency (range 7-30. Higher score is better): number analyzed (Participants) | 36 | 41
  Animal Fluency (range 7-30. Higher score is better) | 16.9 (4.4) | 15.5 (5.6)
  Grooved Pegboard (Range 49-243. Lower score is better): number analyzed (Participants) | 42 | 42
  Grooved Pegboard (Range 49-243. Lower score is better) | 78.0 (20.7) | 77.2 (19.1)

2. Secondary Outcome: Change in Raw Test Scores From Standard Battery of Preferred Neuropsychological Tests
Description: Describe the observed change or stability of neuropsychological test scores in patients who underwent laser ablation surgery. Change will be assessed from raw test scores and demographically corrected standardized scores (where available). For this study, tests include Boston Naming, Trails making Test A and Test B, Digit Span, Logical memory test (subtest from Wechsler Memory Scale IV), BVMT--Brief Visuospatial Memory Test, Animal Fluency test, and Grooved Pegboard.
Time Frame: At least six months from baseline assessment.Subjects were analyzed even if they only had 1 test performed. The baseline test information can still be used even if they didn't have follow up testing done.
Population: Subjects who had LITT and completed baseline and follow-up testing
Measure: Count of Participants; unit: Participants
Arm/Group | PENSAR Subjects
Number analyzed (Participants) | 47
Participants
  Number of subjects who saw no change or improvement in Boston Naming Test: number analyzed (Participants) | 27
  Number of subjects who saw no change or improvement in Boston Naming Test | 25
  Number of subjects who saw no change or improvement in Trails Making Test: number analyzed (Participants) | 34
  Number of subjects who saw no change or improvement in Trails Making Test | 24
  Number of subjects with no change or improvement in Wechsler Adult Intelligence 3 Digital Span Test: number analyzed (Participants) | 33
  Number of subjects with no change or improvement in Wechsler Adult Intelligence 3 Digital Span Test | 30
  Number of subjects who saw no change or improvement in Logical Memory Test: number analyzed (Participants) | 19
  Number of subjects who saw no change or improvement in Logical Memory Test | 19
  Number of subjects who saw no change or improvement in Brief Visiospatial Memory Test: number analyzed (Participants) | 33
  Number of subjects who saw no change or improvement in Brief Visiospatial Memory Test | 29
  Number of subjects who saw no change or improvement in Animal Fluency Test: number analyzed (Participants) | 35
  Number of subjects who saw no change or improvement in Animal Fluency Test | 23
  Number of subjects who saw no change or improvement in Grooved Pegboard Test: number analyzed (Participants) | 37
  Number of subjects who saw no change or improvement in Grooved Pegboard Test | 29

ADVERSE EVENTS:
Time Frame: Baseline testing can occur any time prior to LITT. Follow-up testing occurs at least 6 months after LITT
Description: No adverse events are collected for the PENSAR study.
Arm/Group | PENSAR Subjects
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT05075850/Prot_001.pdf
  • Statistical Analysis Plan (2021-08-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT05075850/SAP_002.pdf